CLINICAL TRIAL: NCT01061840
Title: Phase I Trial of Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Vaccine for Advanced Cancer
Brief Title: Trial of Bi-shRNA-furin and GMCSF Augmented Autologous Tumor Cell Vaccine for Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL-101
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Ewings Sarcoma; Non Small Cell Lung Cancer; Liver Cancer
Keywords: Ewings Sarcoma; Non Small Cell Lung Cancer; Liver Cancer
MeSH Terms: conditions — Sarcoma, Ewing; Carcinoma, Non-Small-Cell Lung; Liver Neoplasms | interventions — FANG vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 x 10 ^7 cells/injection (Experimental): Vigil™
  Interventions: Biological: Vigil™
- 2.5 x 10 ^7 cells/injection (Experimental): Vigil™
  Interventions: Biological: Vigil™
- 1 x 10^6 or 4 x 10^6 cells/injection (Experimental): Vigil™
  Interventions: Biological: Vigil™

INTERVENTIONS:
Biological: Vigil™ — Patients will be treated once a month as long as sufficient material is available for up to 12 doses
  Other Names: bi-shRNAfurin and GMCSF Augmented Autologous Tumor; Cell Vaccine; formerly known as FANG™ Vaccine
  Arms: 1 x 10 ^7 cells/injection
Biological: Vigil™ — Patients will be treated once a month as long as sufficient material is available for up to 12 doses
  Other Names: bi-shRNAfurin and GMCSF Augmented Autologous Tumor; Cell Vaccine; formerly known as FANG™ Vaccine
  Arms: 2.5 x 10 ^7 cells/injection
Biological: Vigil™ — Patients will be treated once a month as long as sufficient material is available for up to 12 doses
  Other Names: bi-shRNAfurin and GMCSF Augmented Autologous Tumor; Cell Vaccine; formerly known as FANG™ Vaccine
  Arms: 1 x 10^6 or 4 x 10^6 cells/injection

SUMMARY:
Autologous Vigil™ vaccine expresses rhGMCSF and bi-shRNAfurin from the Vigil™ plasmid. The GMCSF protein is a potent stimulator of the immune system, recruiting immune effectors to the site of intradermal injection and promoting antigen presentation. The furin bifunctional shRNA blocks furin protein production at the post transcriptional and translational levels. This decrease in furin in turn decreases the conversion of the proforms TGFβ1 and TGFβ2 proteins. Also, reduced furin protein levels have a negative feedback inhibition on TGFβ1 and TGFβ2 gene expression, decreasing the levels of their mRNAs. The resulting decrease in TGFβ1 and TGFβ2 proteins reduces the local immunosuppression they cause and promotes tumor surface antigen and MHC protein display.

DETAILED DESCRIPTION:
Preliminary studies with a variety of vaccines suggest target accessibility (potential immunogenicity) in a variety of solid tumors to immune directed approaches. In an effort to overcome limitations of immunostimulatory cancer vaccines, we have designed a novel autologous vaccine to address inability to fully identify cancer associated antigens, antigen recognition by the immune system (i.e. antigen to immunogen), effector potency, and cancer-induced resistance. We have completed clinical investigations using two different gene vaccine approaches to induce enhancement of tumor antigen recognition which have demonstrated therapeutic efficacy. Specifically, both the use of a GMCSF gene transduced vaccine (GVAX®) and a TGFβ2 antisense gene vaccine (Lucanix®), in separate trials, have demonstrated similar beneficial effects without any evidence of significant toxicity in advanced cancer patients. The GMCSF transgene directly stimulates increased expression of tumor antigen(s) and enhances dendritic cell migration to the vaccination site. TGFβ2 blockade following intracellular TGFβ2 antisense gene expression reduces production of immune inhibiting activity at the vaccine site. This appears to be one of the primary mechanisms of inhibition of immune responsiveness in glioblastoma and lung cancer. In a subsequent Phase I trial we combined both active principles in one autologous vaccine, TAG. TAG vaccine has an excellent safety profile in the first nineteen patients treated (enrollment open to any solid tumor) with one documented CR (melanoma). However, TGFβ1 is the dominant TGFβ family inhibitory effector in the majority of other solid tumors. We describe a unique method of inhibiting both TGFβ1 and TGFβ2 through RNA interference with Furin. We will harvest autologous cancer cells from patients with advanced refractory cancer. We have constructed a bi-shRNAfurin / GMCSF (Vigil™) expression vector plasmid and have successfully demonstrated preclinical activity of the vector function following transfection by electroporation and irradiation of ex vivo autologous tumor cells.

ELIGIBILITY:
Tissue Procurement Inclusion Criteria:

1. Presumptive or histologically confirmed advanced or metastatic non-curable solid tumor (if limited to a single lesion, and may not be a candidate for curative surgery or radiation therapy).
2. For the purpose of the Pediatric study patients with histologic diagnosis of ESFT including: Ewing's sarcoma or primitive neuroectodermal tumor (malignant neuroepithelioma) of the bone or soft tissues, Askin's tumor of the chest and with central nervous system tumors are eligible.
3. Patients with recurrent or refractory ESFT. Patients with de novo poor prognosis/high risk ESFT: (Eligible for vaccine manufacturing at diagnosis but ONLY ELIGIBLE FOR IMMUNOTHERAPY IF DEMONSTRATES PERSISTENT/RECURRENT/ REFRACTORY DISEASE)

   1. Large tumors > 8 cm
   2. Pelvic osseous tumors ANY SIZE
   3. Bilateral pulmonary metastasis
   4. >2 unilateral pulmonary metastasis
4. Clinically (medically) indicated procedure (i.e. biopsy of lesions of recurrent disease, palliative management via resection, thoracentesis, etc.) to collect tumor in sufficient quantity ("golf ball size" estimated weight 10-30 grams, pleural, and/or ascites fluid estimated volume ≥ 500 mL) for vaccine processing.
5. For ESFT patients age ≥12 years.
6. Age ≥18 years (non-ESFT candidates) ECOG performance status (PS) 0-1. Pediatric patients with Lansky or Karnofsky Performance Status Scale ≥ of 50%.
7. Estimated >4 months survival probability.
8. Ability to understand and the willingness to sign a written informed consent document. Pediatric patients must sign an assent with a parent or legal guardian sign a written informed consent.

Inclusion Criteria:

1. Histologically confirmed advanced or metastatic non-curable solid tumor (if limited to a single lesion may not be a candidate for curative surgery or radiation therapy). Successful vaccine manufacture has resulted from tissue/fluid obtained from the following major organ systems: digestive, endocrine, reproductive, respiratory, and urinary.Individuals manufactured under CL-PTL 105 (Phase II Ovarian) may be eligible for enrollment without advanced or metastatic disease.
2. Patients with well differentiated thyroid cancer are eligible for protocol as follows:

   1. Surgically unresectable locally recurrent disease and/or metastatic disease following RAI ablation (if locally recurrent and ultrasound (US) positive, baseline FDG-PET or MRI will be obtained).
   2. Patients with microscopic and/or gross extra thyroidal disease extension without RAI uptake but with a) FDG-PET positive disease or b) suppressed thyroglobulin >1 ng/mL or c) stimulated thyroglobulin >10 ng/L.
   3. Patients with tracheal/esophageal involvement. High mitotic activity or necrosis in pathology does not exclude from the study.

   Note: in Categories a and b, patients can be followed using US locally in addition to standard diagnostic followup menu but, if US only is positive, a FDG-PET or MRI will be obtained. If negative, a rising thyroglobulin titer is required in which case response will be monitored by continued US and suppressed and/or stimulated thyroglobulin. Thyroglobulin titer cannot be used if anti-thyroglobulin antibodies are present).
3. Completed all acceptable therapies with curative intent that are the current standard of care for their respective diseases. If no conventional therapy available, patient may participate after review by sponsor.
4. Recovered from all clinically relevant toxicities related to prior therapies
5. Patients will be allowed to participate following single prior CNS treatment with stereotactic radiotherapy whole brain irradiation and stable without steroid requirement for ≥2 months or following ≥2 prior CNS treatments with stereotactic radiotherapy whole brain irradiation and stable without steroid requirement for ≥4 months.
6. For ESFT patients age ≥12 years.
7. Age ≥18 years (non-ESFT candidates)
8. ECOG performance status (PS) 0-1.Pediatric patients with Lansky or Karnofsky Performance Status Scale ≥ of 50%.
9. Estimated >4 month survival probability.
10. Normal organ and marrow function as defined below:

    Absolute granulocyte count ≥ 1,500/mm3 Absolute lymphocyte count ≥ 500/mm3 Platelets ≥ 100,000/mm3 Total bilirubin ≤2 mg/dL AST(SGOT)/ALT(SGPT) <2x institutional upper limit of normal Creatinine <1.5 mg/dL
11. Ability to understand and the willingness to sign a written informed consent document. Pediatric patients must sign an assent with a parent or legal guardian sign a written informed consent.
12. Negative pregnancy test.
13. Patients must be off all "statin" drugs for ≥2 weeks prior to initiation of therapy.

Exclusion Criteria:

1. Surgery involving general anesthesia, radiotherapy, steroid therapy, or immunotherapy within 4 weeks prior to vaccination. Chemotherapy within 3 weeks prior to entering the study. Palliative radiotherapy is allowable. Collection of lumenal tissue for vaccine manufacture must be avoided.
2. Patients must not have received any other investigational agents within 30 days prior to vaccination.
3. Concurrent tumor-specific hormonal therapy or antiestrogens. (Individuals manufactured under CL-PTL 105 (Phase II Ovarian) are not subject to this exclusion).
4. Patients with known active or symptomatic brain metastases prior to vaccination.
5. Patients with compromised pulmonary disease.
6. Short term (<30 days) concurrent systemic steroids ≤0.25 mg/kg prednisone per day (maximum 7.5 mg/day) and bronchodilators (inhaled steroids) are permitted; other steroid regimens and/or immunosuppressives are excluded while receiving vaccine. Patients requiring steroids following previous CNS radiation for metastatic disease are excluded.
7. Prior splenectomy unless Howell-Jolly bodies are absent.
8. Prior malignancy (excluding nonmelanoma carcinomas of the skin) unless in remission for 2 years.
9. Kaposi's Sarcoma.
10. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Patients who are pregnant or nursing.
12. Patients with known HIV.
13. Patients with chronic Hepatitis B and C infection. For patients with hepatocellular carcinoma (HCC), the presence of chronic HBV and HCV is NOT an exclusion. Patients must have a viral titer <50 IU/ml x 2 at a minimum of 2 weeks apart.
14. Patients with uncontrolled autoimmune diseases.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
To determine safety following the administration of bi-shRNAfurin and GMCSF autologous tumor cell (Vigil™) vaccine in advanced solid tumor patients who have no acceptable form of standard therapy with curative intent. | Participants will be followed for life

SECONDARY OUTCOMES:
To determine time to progression. To evaluate the effect of Vigil™ vaccine on immune stimulation. To evaluate whether lower cell doses would activate ELISPOT responses and to compare durability of dose elicited responses. | Participants will be followed for life.

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Centers
Locations (4):
- United States (4):
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Dartmouth-Hitchcock Medical Center/ Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Cancer Care Northwest, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nemunaitis J, Barve M, Orr D, Kuhn J, Magee M, Lamont J, Bedell C, Wallraven G, Pappen BO, Roth A, Horvath S, Nemunaitis D, Kumar P, Maples PB, Senzer N. Summary of bi-shRNA/GM-CSF augmented autologous tumor cell immunotherapy (FANG) in advanced cancer of the liver. Oncology. 2014;87(1):21-9. doi: 10.1159/000360993. Epub 2014 Jun 25. PMID 24968881
- [Result] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Result] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Result] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Result] Oh J, Barve M, Senzer N, Aaron P, Manning L, Wallraven G, Bognar E, Stanbery L, Horvath S, Manley M, Nemunaitis J, Walter A, Rocconi RP. Long-term follow-up of Phase 2A trial results involving advanced ovarian cancer patients treated with Vigil(R) in frontline maintenance. Gynecol Oncol Rep. 2020 Sep 17;34:100648. doi: 10.1016/j.gore.2020.100648. eCollection 2020 Nov. No abstract available. PMID 33364285
- [Result] Rocconi RP, Stanbery L, Madeira da Silva L, Barrington RA, Aaron P, Manning L, Horvath S, Wallraven G, Bognar E, Walter A, Nemunaitis J. Long-Term Follow-Up of Gemogenovatucel-T (Vigil) Survival and Molecular Signals of Immune Response in Recurrent Ovarian Cancer. Vaccines (Basel). 2021 Aug 12;9(8):894. doi: 10.3390/vaccines9080894. PMID 34452019